CLINICAL TRIAL: NCT05161546
Title: Study of Bipolar Disorders and Retinal Electrophysiological Markers
Acronym: BIMAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Malfunctions of the Retinaute® but no adverse effects on participants. Study interrupted for BioSerenity to make technical corrections. Long immobilization of the device and conditions for reusing it not adapted to the continuation of the study.
Sponsor: Centre Psychothérapique de Nancy (Other)
Collaborators: BioSerenity (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RIPH 2021-03; IDRCB 2021-A01644-37 (Other: ANSM)
Record Dates: First submitted 2021-09-28; First posted 2021-12-17 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; biomarker; electroretinogram; electroencephalogram; neurocognition; actigraphy; retina
MeSH Terms: conditions — Bipolar Disorder | interventions — Electroencephalography; Actigraphy; Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: The BiMAR study is an open-label and non-randomized comparative monocentric study applied in psychiatry and neuroscience.
  This research included two groups of adult subjects: a group of patients with BD in the euthymic phase and a group of healthy control subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with bipolar disorder (BD) (Experimental): Electrophysiological recordings with ERG and EEG will be performed with a virtual reality headset after a standardized clinical evaluation (first visit).
  Then, an actigraphic monitoring of 21 consecutive days will be carried out. At the end of this period a neuropsychological evaluation will be performed during a second visit.
  Between day 23 and day 28 (after the second visit), patients will be offered to assess the retinal structure and microvascularization using Spectral Domain Optical Coherence Tomography (SD-OCT) and OCT-Angiography (OCT-A).
  Interventions: Device: EEG and ERG measurements (Retinaute®, BioSerenity); Device: Actigraphy (Motion Watch 8®, CamNtech); Behavioral: Neuropsychological assessments; Device: Optical Coherence Tomography (OCT)
- healthy volunteers (Active Comparator): Electrophysiological recordings with ERG and EEG will be performed with a virtual reality headset after a standardized clinical evaluation (first visit).
  Then, an actigraphic monitoring of 21 consecutive days will be carried out. At the end of this period a neuropsychological evaluation will be performed during a second visit.
  Interventions: Device: EEG and ERG measurements (Retinaute®, BioSerenity); Device: Actigraphy (Motion Watch 8®, CamNtech); Behavioral: Neuropsychological assessments

INTERVENTIONS:
Device: EEG and ERG measurements (Retinaute®, BioSerenity) — The Retinaute® is a portable medical device developed by BioSerenity, France, for performing flash and pattern ERG. It comes in the form of a virtual reality headset, which can be used in outpatient facilities. It is non-invasive and uses skin electrodes for the collection of parameters.
  ERG signals will be supplemented with 4 EEG channels, via cup electrodes applied to the skull and allowing the concomitant performance of an EEG.
Device: Actigraphy (Motion Watch 8®, CamNtech) — Actigraphy is an ecological and non-invasive method allowing a reliable characterization of the sleep/wake cycle. It is a portable system for continuously measuring the motor activity of an individual and appreciating the alternation of activity periods (wakefulness) and rest periods (sleep).
  An actigraph (MotionWatch8®, CamNtech) looks like a wristwatch that will be worn continuously, by convention on the wrist of the non-dominant hand, over periods ranging from several days to several weeks (here 21 days). Actigraphy does not present a known risk.
Behavioral: Neuropsychological assessments — The purpose of this assessment is to establish a cognitive profile for each participant. It uses a series of tests widely described in the literature and commonly used today.
Device: Optical Coherence Tomography (OCT) — The Spectral Domain Optical Coherence Tomography (SD-OCT) is a modern ocular imaging process using infrared radiation and allowing to obtain in a few seconds, and in a non-invasive way, images in section of the eye. The OCT-Angiography (OCT-A) module increments on the OCT. It can detect the movement of the blood elements from sequential SD-OCT slices taken at the same location of the retina and obtain a map of the retinal and choroidal vessels, without injection of fluorescent dye. The device used for both exams will be the OCT spectral RS 3000 Advance 2 + Angioscan (NIDEK, Gamagori, Japan). SD-OCT and OCT-A examinations are fast, painless, non-contact and last less than a minute. There is no particular risk.
  Arms: patients with bipolar disorder (BD)

SUMMARY:
The BIMAR study aims to compare electrophysiological data measured with electroretinogram (ERG) and electroencephalogram (EEG) between a group of euthymic patients with bipolar disorder (BD) and a group of healthy controls subjects.

Secondarily, the investigators also want to:

* Compare combined electrophysiological measurements with ERG and EEG between the two groups.
* Identify relations between clinical, neuropsychological and circadian phenotypes in patients with BD and electrophysiological measurements measured with ERG and EEG.

The main hypothesis of the investigators is that differences exist in the ERG and EEG measurements between subjects with BD and healthy subjects. Those differences could be identified as candidate markers for BD which, if confirmed in later studies, could be used in current practice to guide the management of patients with BD.

DETAILED DESCRIPTION:
Bipolar disorders (BD) is a common, chronic and disabling psychiatric condition. In addition to being characterized by significant clinical heterogeneity, notable disturbances of sleep and cognitive function are frequently observed in all phases of the disease. Currently, there is no readily available biomarker in current clinical practice to help diagnose or predict the disease course. Thus, identification of biomarkers in BD is today a major challenge. In this context, the study of electrophysiological biomarkers based on electroretinogram (ERG) and electroencephalogram (EEG) measurements in BD seems highly promising. The BiMAR study aims to compare electrophysiological data measured with ERG and EEG between a group of euthymic patients with BD and a group of healthy control subjects. Secondarily, the investigators will also describe the existing potential relationship between clinical, sleep and neuropsychological phenotypes of patients and electrophysiological data.

The BiMAR study is a comparative and monocentric study carried out at the Expert Center for BD in Nancy, France. In total, 70 euthymic adult patients with BD and 70 healthy control subjects will be recruited. Electrophysiological recordings with ERG and EEG will be performed with a virtual reality headset after a standardized clinical evaluation to all participants. Then, an actigraphic monitoring of 21 consecutive days will be carried out. At the end of this period a neuropsychological evaluation will be performed during a second visit. The primary outcome will be electrophysiological measurements with ERG flash and pattern. Secondary outcomes will be EEG data, sleep settings, clinical and neuropsychological assessments. For patients only, a complementary ancillary study, carried out at the University Hospital of Nancy, will be proposed to assess the retinal structure and microvascularization using Optical Coherence Tomography. Recruitment will begin in December 2021 and will continue until the end of June 2023.

The BiMAR study will contribute to identifying candidate ERG electrophysiological markers for helping the diagnosis of BD and identify subgroups of patients with different clinical profiles. Eventually, this would allow earlier diagnosis and personalized therapeutic interventions.

ELIGIBILITY:
Inclusion criteria :

1. Patients:

   * been diagnosed with BD according to the Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV) diagnostic criteria using the Mini International Neuropsychiatric Interview (MINI)
   * currently euthymic for at least 3 months prior to the study, as defined by a score below 10 on the Montgomery-Asberg Depression Rating Scale (MADRS) which assesses depression and by a score below 8 on the Young Mania Rating Scale (YMRS) which assesses mania
   * age 18 or more
2. Healthy volunteers:

   * not suffer from a personal psychiatric pathology verified with the MINI
   * age 18 or more

Exclusion criteria for all participants (patients and healthy volunteers):

* suffer from psychiatric pathology or substance use disorders according to DSM-IV criteria measured with the MINI, excluding BD for the patient group
* suffer from neurological or retinal pathology
* having a shift work or a get-lag in the last 15 days
* criteria incompatible with the use of the virtual reality headset (Retinaute®,BioSerenity) like having an allergy to one of the components of the textile
* persons treated by sismotherapy during the past year
* persons with an uncorrected visual impairment or disabling hearing impairment that does not allow neuropsychological tests to be performed
* subjects with an intellectual disability making it difficult to participate in the study or to understand and follow informations provided to them
* adults legally protected
* pregnant or breastfeeding women
* subjects already participating in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Modification of amplitude measured with flash and pattern electroretinogram | Day 0 (=day of inclusion)
  amplitude in microvolt
Modification of implicite time measured with flash and pattern electroretinogram | Day 0 (=day of inclusion)
  implicite time in millisecond

SECONDARY OUTCOMES:
Modification of amplitude measured with electroencephalogram | Day 0 (=day of inclusion)
  amplitude of the P100, N170 and N200 waves amplitude in microvolt
Modification of latency measured with electroencephalogram | Day 0 (=day of inclusion)
  latency of the P100, N170 and N200 waves latency in millisecond
Actigraphy | from Day1 to Day21
  evaluation of sleep/wake cycles
Sleep diary | from Day 1 to Day 21
  self reported tool of sleeping and waking times
Visual Object and Space Perception battery (VOSP) | visit n ° 2 (=between Day 22 and Day 27)
  test of visual cognition
California Verbal Learning Test (CVLT) | visit n ° 2 (=between Day 22 and Day 27)
  assessment of verbal episodic memory
Continuous Performance Task (CPT-III) | visit n ° 2 (=between Day22 and Day27)
  test of sustained attention
Verbal Fluency Task | visit n ° 2 (=between Day 22 and Day 27)
  test of verbal functioning
Test of Attention Assessment (TAP) | visit n ° 2 (=between Day 22 and Day 27)
  test of attentional performance
Montreal Cognitive Assessment (MoCA) | visit n ° 2 (=between Day 22 and Day 27)
  screening assessment for detecting cognitive impairment

OTHER OUTCOMES:
Mini International Neuropsychiatric Interview (MINI) | Day 0 (=day of inclusion)
  questionnaire to diagnose psychiatric disorders
Montgomery-Asberg Depression Rating Scale (MADRS) | Day 0 (=day of inclusion)
  rating scale measuring depressive symptoms
Montgomery-Asberg Depression Rating Scale (MADRS) | at the visit n ° 2 (=between Day 22 and Day 27)
  rating scale measuring depressive symptoms
Young Mania Rating Scale (YMRS) | Day 0 (=day of inclusion)
  rating scale measuring manic symptoms
Young Mania Rating Scale (YMRS) | at the visit n ° 2 (=between Day 22 and Day 27)
  rating scale measuring manic symptoms
Pittsburgh Sleep Quality Index (PSQI) | Day 0 (=day of inclusion)
  assess the subjective quality of sleep during the past month
Pittsburgh Sleep Quality Index (PSQI) | at the visit n ° 2 (=between Day 22 and Day 27)
  assess the subjective quality of sleep during the past month
Insomnia Severity Index (ISI) | Day 0 (=day of inclusion)
  assess the severity of insomnia
Insomnia Severity Index (ISI) | at the visit n ° 2 (=between Day 22 and Day 27)
  assess the severity of insomnia
Epworth sleepiness scale (ESS) | Day 0 (=day of inclusion)
  assess the daytime sleepiness
Epworth sleepiness scale (ESS) | at the visit n ° 2 (=between Day 22 and Day 27)
  assess the daytime sleepiness
Horne and Ostberg circadian typology questionnaire | Day 0 (=day of inclusion)
  assess the circadian rhythm type by evaluating the daily sleep-wake habits and the times of day when certain activities are performed with preferences
Horne and Ostberg circadian typology questionnaire | at the visit n ° 2 (=between Day 22 and Day 27)
  assess the circadian rhythm type by evaluating the daily sleep-wake habits and the times of day when certain activities are performed with preferences
Composite Scale of Morningness (CSM) | Day 0 (=day of inclusion)
  measure of behavioral temporal preference
Composite Scale of Morningness (CSM) | at the visit n ° 2 (=between Day 22 and Day 27)
  measure of behavioral temporal preference
Circadian Type Inventory (CTI) | Day 0 (=day of inclusion)
  assess of amplitude and stability of rhythms
Circadian Type Inventory (CTI) | at the visit n ° 2 (=between Day 22 and Day 27)
  assess of amplitude and stability of rhythms
The Berlin Questionnaire | Day 0 (=day of inclusion)
  estimate the risk of Obstructive Sleep Apnea syndrome
The Berlin Questionnaire | at the visit n ° 2 (=between Day 22 and Day 27)
  estimate the risk of Obstructive Sleep Apnea syndrome
Quick Inventory of Depressive Symptomatology self-report (QIDS-SR) | Day 0 (=day of inclusion)
  self reported rating scale measuring depressive symptoms
Altman Self-Rating Mania Scale (ALTMAN) | Day 0 (=day of inclusion)
  self reported rating scale measuring manic symptoms
State Trait Inventory Anxiety (STAI-A) | Day 0 (=day of inclusion)
  self reported rating scale measuring anxiety symptoms
Multidimensional Assessment of Thymic States (MATHYS) | Day 0 (=day of inclusion)
  self reported assessment of emotional reactivity
Patient Rated Inventory of Side Effects (PRISE-M) | Day 0 (=day of inclusion)
  self reported assessment of tolerance to treatments
Medication Adherence Rating (MARS) | Day 0 (=day of inclusion)
  self reported assessment of adherence to treatments
Alda Scale | Day 0 (=day of inclusion)
  assess response to lithium treatment
Functioning Assessment Short Test (FAST) | Day 0 (=day of inclusion)
  assess patient's functioning
Clinical Global Impression Scale (CGI) | Day 0 (=day of inclusion)
  assess patient's functioning
Affective Instability Measure (AIM) | Day 0 (=day of inclusion)
  assess oscillations of intense affect
Affective Lability Scale (ALS) | Day 0 (=day of inclusion)
  assess the emotional lability
Buss-Durkee Hostility Inventory (BDHI) | Day 0 (=day of inclusion)
  assess the hostility
Barrat Impulsivity Scale (BIS-10) | Day 0 (=day of inclusion)
  assess the impulsivity
Wender Utah Rating Scale (WURS) | Day 0 (=day of inclusion)
  check for a history of attention deficit hyperactivity disorder
Childhood Trauma Questionnaire (CTQ) | Day 0 (=day of inclusion)
  check for trauma in childhood
Fagerström test | Day 0 (=day of inclusion)
  assess the tobacco addiction
Edinburgh Handedness Inventory | Day 0 (=day of inclusion)
  assess the manual preference
Spectral Domain Optical Coherence Tomography (SD-OCT) | between Day 23 and Day 28
  evaluation of retinal structure
Optical Coherence Tomography Angiography (OCT-A) | between Day 23 and Day 28
  evaluation of retinal vascularity

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SCHWITZER, MD, PhD, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapique de Nancy, Laxou, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwitzer T, Schwan R, Bubl E, Lalanne L, Angioi-Duprez K, Laprevote V. Looking into the brain through the retinal ganglion cells in psychiatric disorders: A review of evidences. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Jun 2;76:155-162. doi: 10.1016/j.pnpbp.2017.03.008. Epub 2017 Mar 20. PMID 28336492
- [Background] Tan A, Schwitzer T, Conart JB, Angioi-Duprez K. Study of retinal structure and function in patients with major depressive disorder, bipolar disorder or schizophrenia: A review of the literature. J Fr Ophtalmol. 2020 May;43(5):e157-e166. doi: 10.1016/j.jfo.2020.04.004. Epub 2020 May 4. PMID 32381369
- [Background] Hebert M, Merette C, Gagne AM, Paccalet T, Moreau I, Lavoie J, Maziade M. The Electroretinogram May Differentiate Schizophrenia From Bipolar Disorder. Biol Psychiatry. 2020 Feb 1;87(3):263-270. doi: 10.1016/j.biopsych.2019.06.014. Epub 2019 Jun 27. PMID 31443935
- [Derived] Gross G, Tursini K, Albuisson E, Angioi-Duprez K, Conart JB, Louis Dorr V, Schwan R, Schwitzer T. Bipolar disorders and retinal electrophysiological markers (BiMAR): Study protocol for a comparison of electroretinogram measurements between subjects with bipolar disorder and a healthy control group. Front Psychiatry. 2022 Sep 8;13:960512. doi: 10.3389/fpsyt.2022.960512. eCollection 2022. PMID 36159928